CLINICAL TRIAL: NCT03079635
Title: The Effect of Breakfast Intake on Energy Expenditure and Hunger in Young Women
Brief Title: Breakfast and Energy Expenditure in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-09-124
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight (Active Comparator): This group will be administered two breakfast beverages with a one- to two-week washout period between beverages. The beverages will be a control or an isocaloric, macronutrient matched breakfast beverage with omega-3 fatty acids.
  Interventions: Dietary Supplement: Control; Dietary Supplement: Omega 3 fatty acids
- Overweight and Obese (Active Comparator): This group will be administered two breakfast beverages with a one- to two-week washout period between beverages. The beverages will be a control or an isocaloric, macronutrient matched breakfast beverage with omega-3 fatty acids.
  Interventions: Dietary Supplement: Control; Dietary Supplement: Omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: Control — Beverage provided and a four hour postprandial assessment of energy metabolism using a metabolic cart and appetite using a visual analog scale follows.
Dietary Supplement: Omega 3 fatty acids — Beverage provided and a four hour postprandial assessment of energy metabolism using a metabolic cart and appetite using a visual analog scale follows.

SUMMARY:
The purpose of this research is to determine if body composition influence the effect of breakfast composition on postprandial (post-meal) hunger, metabolic and energy expenditure response in normal weight, overweight, and obese young women.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 18.5
* No medication

Exclusion Criteria:

* Food allergies
* Habitual breakfast skipping (> 5 times per week)
* Picky eater
* Dietary restrictions

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Energy metabolism/expenditure | Four hours
  Energy expenditure and thermic effect of feeding will be measured using a TrueMax 2400 metabolic cart

SECONDARY OUTCOMES:
Appetite | Four hours
  Postprandial appetite will be assessed using visual analog scales

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No